CLINICAL TRIAL: NCT04615416
Title: Open Trial of Emotion Regulation Training Via Telehealth for Distressed Adults During the COVID-19 Pandemic
Brief Title: Emotion Regulation Training Via Telehealth During the COVID-19 Pandemic
Acronym: ERT-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Douglas Mennin, Professor of Clinical Psychology, Teachers College, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-269
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Distress, Emotional; Emotional Dysfunction; Anxiety; Depression
Keywords: Emotion Regulation; Distress Disorders; Anxiety; Depression; COVID-19 Pandemic; Telehealth
MeSH Terms: conditions — Anxiety Disorders; Depression; Emotional Regulation; COVID-19

STUDY DESIGN:
Intervention Model Description: All participants will receive a 9-session version of Emotion Regulation Training delivered semi-weekly via synchronous telehealth using videoconferencing software and an asynchronous Internet-based Online platform to supplement the content covered in each session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Emotion Regulation Training via Telehealth (Experimental): All participants will receive 9 sessions of Emotion Regulation Training delivered via telehealth. These individualized therapy sessions are 1-hour in length and occur semi-weekly over the course of four weeks.
  Interventions: Behavioral: Emotion Regulation Training via Telehealth

INTERVENTIONS:
Behavioral: Emotion Regulation Training via Telehealth — The initial stage of treatment focuses on psychoeducation about anxiety/depression, the impact that these cognitions/behaviors/emotions have on recent situations, and self-monitoring of worry/anxiety/depression. The sessions focus on the development of skills that help understand and regulate one's emotional experience (i.e., recognizing emotions when they are happening, identifying the meaning of a given emotion experience, soothing oneself in the context of negative emotional experiences). Following the development of these skills, sessions focus on the application of somatic awareness and emotion regulation skills while imagining emotionally evocative themes. The remaining session focuses on terminating therapy, relapse prevention, and future goals. An Internet-based online platform will be used to promote engagement with and increase accessibility to between-session skills practice and treatment-related activities (e.g., self-monitoring, session summaries, worksheets).
  Other Names: Emotion Regulation Therapy (ERT)

SUMMARY:
This study is an open trial designed specifically to address the need for evidence-based treatment delivered via telehealth to individuals that are currently struggling with mental health issues during the COVID-19 pandemic, with the overarching goal of helping residents of New York adversely impacted by the pandemic to effectively manage their anxiety, stress, and depression during this unprecedented time in human history.

DETAILED DESCRIPTION:
The present study is evaluating whether this ERT treatment program delivered via telehealth demonstrates efficacy in: 1) reducing symptoms of psychological distress (e.g., anxiety, depression, worry, rumination); 2) improving outcomes specific to the ERT mechanism-based model (e.g., attentional control, decentering, reappraisal); 3) improving quality of life and functioning, for adults aged 18-65 years old.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years during the time of participation
* Endorses distress and worry/rumination exacerbated by the COVID-19 pandemic
* Access to a mobile device (e.g., smartphone, personal computer, laptop, tablet) connected to the Internet

Exclusion Criteria:

* Active suicidal intent
* Current substance dependence disorder (within the past year)
* Current or past psychotic disorder, Bipolar-I disorder, or dementia
* Primary DSM-5 diagnosis of borderline or narcissistic personality disorder
* Currently receiving any other form of psychosocial treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Changes in Anxiety, Depression, and Distress: Mood and Anxiety Symptoms Questionnaire (MASQ) | Pre-Treatment, Post-Treatment (4-5 weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Scale = 1-5 (minimum = 30; maximum = 150; higher scores indicate worse outcomes)
Changes in Anxiety, Depression, and Distress: Depression Anxiety Stress Scale (DASS) | Pre-Treatment, Post-Treatment (4-5 weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Scale = 0-4 (minimum = 0; maximum = 84; higher scores indicate worse outcomes)
Changes in Worry: Penn State Worry Questionnaire (PSWQ) | Pre-Treatment, Post-Treatment (4-5 weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Scale = 1-5 (minimum = 12; maximum = 60; higher scores indicate worse outcomes)
Changes in Rumination: Rumination-Reflection Questionnaire (RRQ) | Pre-Treatment, Post-Treatment (4-5 weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Scale = 1-5 (minimum = 12; maximum = 60; higher scores indicate worse outcomes)
Changes in Functional Impairment: Sheehan Disability Scale (SDS) | Pre-Treatment, Post-Treatment (4-5 weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Scale = 0-10 (minimum = 0; maximum = 30; higher scores indicate worse outcomes)
Changes in Life Satisfaction: Brief Multidimensional Students' Life Satisfaction Scale (BMSLSS) | Pre-Treatment, Post-Treatment (4-5 weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Scale = 1-6 (minimum = 5; maximum = 30; higher scores indicate better outcomes)
Changes in Life Satisfaction: Patient-Reported Outcomes Measurement Information System (PROMIS): Meaning and Purpose | Pre-Treatment, Post-Treatment (4-5 weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Scale = 1-5 (minimum = 4; maximum = 20; higher scores indicate better outcomes)

SECONDARY OUTCOMES:
Semi-Weekly Measures of Treatment Changes in Anxiety: Patient-Reported Outcomes Measurement Information System (PROMIS): Anxiety | Semi-weekly over the course of four weeks
  Scale = 1-5 (minimum = 4; maximum = 20; higher scores indicate worse outcomes)
Semi-Weekly Measures of Treatment Changes in Depression: Patient-Reported Outcomes Measurement Information System (PROMIS): Depression | Semi-weekly over the course of four weeks
  Scale = 1-5 (minimum = 4; maximum = 20; higher scores indicate worse outcomes)
Semi-Weekly Measures of Treatment Changes in Depression Symptoms | Semi-weekly over the course of four weeks
  Quick Inventory of Depressive Symptoms(QUIDS)
Semi-Weekly Measures of Treatment Changes in Distress | Semi-weekly over the course of four weeks
  Distress Thermometer (DT)
Semi-Weekly Measures of Treatment Changes in Worry: Brief Penn State Worry Questionnaire (PSWQ) | Semi-weekly over the course of four weeks
  Scale: 1-5 (minimum = 3; maximum = 15; higher scores indicate worse outcomes)
Semi-Weekly Measures of Treatment Changes in Rumination: Brief Rumination-Reflection Questionnaire (RRQ) | Semi-weekly over the course of four weeks
  Scale = 1-5 (minimum = 3; maximum = 15; higher scores indicate worse outcomes)
Semi-Weekly Measures of Treatment Changes in Metacognitive Regulation: Emotion Regulation Questionnaire (ERQ) | Semi-weekly over the course of four weeks
  Scale = 1-5 (minimum = 6; maximum = 30; higher scores indicate better outcomes)
Semi-Weekly Measures of Treatment Changes in Metacognitive Regulation: Experiences Questionnaire (EQ) | Semi-weekly over the course of four weeks
  Scale = 1-5 (minimum = 5; maximum = 25; higher scores indicate better outcomes)
Semi-Weekly Measures of Treatment Changes in Attentional Regulation: The Attentional Control Scale (ACS) | Semi-weekly over the course of four weeks
  Scale = 1-4 (minimum = 6; maximum = 24; higher scores indicate better outcomes)
Satisfaction and Usability of Treatment: Client Satisfaction Questionnaire (CSQ) | Post-Treatment (4-5 weeks after starting treatment)
  Scale = 1-4 (minimum = 4; maximum = 16; higher scores indicate better outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Mennin, Ph.D., Principal Investigator — Teachers College, Columbia University
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mennin DS, Fresco DM, O'Toole MS, Heimberg RG. A randomized controlled trial of emotion regulation therapy for generalized anxiety disorder with and without co-occurring depression. J Consult Clin Psychol. 2018 Mar;86(3):268-281. doi: 10.1037/ccp0000289. PMID 29504794
- [Background] Renna ME, Quintero JM, Soffer A, Pino M, Ader L, Fresco DM, Mennin DS. A Pilot Study of Emotion Regulation Therapy for Generalized Anxiety and Depression: Findings From a Diverse Sample of Young Adults. Behav Ther. 2018 May;49(3):403-418. doi: 10.1016/j.beth.2017.09.001. Epub 2017 Sep 8. PMID 29704969